CLINICAL TRIAL: NCT00900640
Title: Reactions to Contrast Media (CM) Administered at the Time of Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Reactions to Contrast Media (CM) Administered at the Time of the Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: ERCP Contrast 144-09
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Contrast Allergies
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ERCP group: All patients who have been scheduled for an ERCP due to medical necessity will be considered for this study.
  Interventions: Procedure: ERCP as medically indicated by subjects referring physician

INTERVENTIONS:
Procedure: ERCP as medically indicated by subjects referring physician — Determine the incidence of adverse reactions to CM administered during ERCP in patients with prior reaction to IV CM administration and/or shellfish allergy.

SUMMARY:
The aim of this study is to prospectively document the incidence of CM adverse reactions at the time of ERCP and to determine whether various perceived risk factors are predictive of adverse reaction.

Adverse reactions to iodine containing contrast media (CM) have been described after endoscopic retrograde cholangiopancreaticography (ERCP) but have been difficult to study due to their extremely low incidence. Adverse reactions can be classified by severity (mild, moderate or severe) or underlying mechanism (idiosyncratic versus nonidiosyncratic). Nonidiosyncratic reactions are related to the dose and osmolality of the CM; these are not observed during ERCP due to the relative small amount of systemic absorption of CM. Idiosyncratic reactions on the other hand are not dose-dependent and generally occur shortly after administration of CM.

Premedication with corticosteroids, H1/H2 -blockers and the use of low osmolality CM is beneficial in preventing nonidiosyncratic reactions during intravascular administration. However their role in during ERCP is unclear as CM is not injected into the intravascular space. Currently there are no formal recommendations and clinical practice varies considerably. The general purpose of this study is to determine the incidence of CM reactions during ERCP and to determine whether various risk factors are predictive of idiosyncratic reactions. Based on these results, we hope to develop guidelines for the use of prophylaxis to prevent CM reactions in ERCP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Scheduled to undergo ERCP at the University of Florida, Gainesville, FL
3. History of prior reaction to IV CM and/or shellfish allergy
4. Subject must be able to give informed consent

Exclusion Criteria:

1. Any contraindication to performing ERCP.
2. Participation in another research protocol that could interfere or influence the outcomes measures of the present study.
3. The subject is unable/unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who medically need an ERCP to further evaluate or treat their medical condition.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Determine the incidence of adverse reactions to CM administered during ERCP in patients with prior reaction to IV CM administration and/or shellfish allergy. | at the time of the subjects ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Peter V. Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands UF endoscopy Center, Gainesville, Florida, United States